CLINICAL TRIAL: NCT00286234
Title: Niacin, N-3 Fatty Acids and Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Dakota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William S. Harris, PhD, FAHA, FNLA, Professor, University of South Dakota
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK61486 (completed); R01DK061486 (NIH)
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Syndrome; Hypertriglyceridemia
Keywords: triglycerides; HDL-cholesterol; insulin resistance; omega-3 fatty acids; niacin
MeSH Terms: conditions — Metabolic Syndrome; Hypertriglyceridemia; Insulin Resistance | interventions — Omacor; Niacin; Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Dual placebo
  Interventions: Drug: placebo
- 2 (Experimental): niaspan
  Interventions: Drug: extended release niacin
- 3 (Experimental): lovaza
  Interventions: Drug: omega-3 acid ethyl esters
- 4 (Experimental): combined therapy
  Interventions: Drug: combined treatment

INTERVENTIONS:
Drug: omega-3 acid ethyl esters — 4 q qd
  Other Names: lovaza omacor
  Arms: 3
Drug: extended release niacin — 2 g qpm
  Other Names: niaspan
  Arms: 2
Drug: placebo — omacor placebo plus niaspan placebo
  Arms: 1
Drug: omega-3 acid ethyl esters — 4 g qd
  Other Names: lovaza omacor
  Arms: 3
Drug: combined treatment — omega-3 acid ethyl esters 4 g qd and extended release niacin, titrate up to 2 g Qpm
  Other Names: lovaza, omacor; niaspan
  Arms: 4

SUMMARY:
This research study is being conducted to test the effects of two drugs on blood lipids (cholesterol and triglycerides) and blood sugar (glucose) levels in patients with diabetes or "pre-diabetes" (both of which have a condition called "insulin-resistance"). These products are Niaspan (extended release nicotinic acid) and Omacor (omega-3 acid ethyl esters). We hypothesize that the combination of Niaspan and Omacor will reduce serum triglyceride levels, increase HDL-cholesterol levels and do so without altering glucose levels.

DETAILED DESCRIPTION:
The insulin resistance syndrome (IRS) afflicts approximately 25% of the US adult population. Its principal components include some or all of the following: central obesity, elevated triglyceride levels, decreased high density lipoprotein cholesterol (HDL-C) levels, a preponderance of small, dense low density lipoprotein (LDL) particles, hyperglycemia, hypertension, and increased thrombotic tendency. Subjects with the IRS are at increased risk for type 2 diabetes and/or coronary heart disease (CHD). While lifestyle changes (diet and exercise) often improve many of the manifestations of the IRS, pharmacotherapy is often needed to normalize individual components.

In recent studies from our laboratory, niacin and fish oil (n-3 fatty acids, FA) used in combination in insulin resistant individuals led to an expected improved the lipid phenotype (reduced triglycerides, increased HDL-C, and fewer, small, dense LDL particles). What was not expected, however, was that an important marker of adipose tissue insulin resistance - meal-induced suppression of free fatty acid (FFA) flux - would be improved as well. Further, knowing that these agents (given as monotherapy) have been reported to worsen glycemia in diabetic subjects, we were surprised to find no significant deterioration in glycemic control. Further preliminary studies in patients with poorly-controlled type 2 diabetes confirmed the ability of this combination of over-the-counter natural agents to significantly improve the lipid profile without adverse effects on glycemia.

Our working hypothesis is that excessive FFA flux from adipose tissue raises serum triglyceride concentrations and leads to other manifestations of the IRS. FFA flux is chronically elevated in insulin resistant subjects due to the insensitivity (i.e., resistance) of their adipocytes to the anti-lipolytic effects of insulin. Released FFA (especially from visceral adipose depots) stimulate hepatic triglyceride synthesis, leading to elevated serum triglyceride levels which subsequently contribute to reduced HDL-C and increased small, dense LDL concentrations. In addition, a high FFA flux can interfere with whole body glucose disposal. If this hypothesis is true, then interventions that improve adipocyte insulin sensitivity may be expected to improve a spectrum of risk factors associated with the insulin resistant state.

Since our preliminary studies support this hypothesis, we propose the following four specific aims which will be tested in a 4-arm, randomized, placebo-controlled, double blind trial:

Specific Aim 1. To test the hypothesis that n-3 FA and niacin (given singly and in combination) will enhance insulin-mediated suppression of FFA rate of appearance (Ra; a surrogate for adipose tissue insulin sensitivity) in insulin resistant subjects.

Specific Aim 2. To test the hypothesis that n-3 FA and niacin (given singly and in combination) will improve insulin sensitivity in insulin resistant subjects.

Specific Aim 3. To test the hypothesis that n-3 FA and niacin (given singly and in combination) will reduce VLDL-triglyceride production rates in insulin resistant subjects.

Specific Aim 4. To test the hypothesis that n-3 FA and niacin (given singly and in combination) will improve the dyslipidemic profile (i.e., reduce serum triglyceride and small, dense LDL concentrations and elevate HDL-C concentrations) in insulin resistant subjects.

At the completion of these studies, we expect to have detailed information on the potential therapeutic efficacy and the kinetic mechanism of action of combined treatment with n-3 FA and niacin. A better understanding of the action of these agents should lead to a clearer appreciation of the relationship between FFA flux and insulin resistance, to more effective therapy for the dyslipidemia of insulin resistance and ultimately to reduced risk for CAD in this burgeoning patient population.

ELIGIBILITY:
Inclusion Criteria:

40 and 69 years of age Male or female (without hormonal cycling as described below) BMI > 25 Fasting serum triglycerides > 150 mg/dL Ratio of TG/HDL-C > 3.5

Exclusion Criteria:

BMIs > 40 kg/m2 TG > 750 mg/dL HDL-C < 10 mg/dL Presence of other secondary causes of dyslipidemia or hyperglycemia such as hepatic, renal, thyroid or other endocrine diseases History of hypersensitivity to niacin or fish oils History of gout, hepatitis, peptic ulcer or cardiovascular disease Presence of diabetes mellitus, whether controlled by diet or drugs. (We will eliminate subjects with undiagnosed diabetes by screening for fasting glucose > 126 mg/dL) Use of any dietary supplements providing more than 50 mg of niacin or 100 mg of n-3 FA Use of any herbal preparations or weight-loss products Taking any lipid-lowering drugs for at least four weeks prior to screening for the study Medically-required treatment with nitrates, calcium channel blockers, or adrenergic blocking agents (per the Niaspan package insert) Hemoglobin < 12 g/dL (owing to the significant amount of blood being drawn) LDL-C > 145 mg/dL. (This restriction will prevent the randomization of any subject whose LDL-C levels, if assigned to an n-3 FA group, might rise by 10% and thus exceed 160 mg/dL) Known substance abuse Participation in a clinical drug trial anytime during the 30 days prior to screening Anyone whom the investigators judge to be a poor candidate

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Harris, PhD, Principal Investigator — Sanford Research/USD
Locations (1):
- Sanford Clinic Clinical Research Services, Sioux Falls, South Dakota, United States

REFERENCES:
- [Derived] Savinova OV, Fillaus K, Harris WS, Shearer GC. Effects of niacin and omega-3 fatty acids on the apolipoproteins in overweight patients with elevated triglycerides and reduced HDL cholesterol. Atherosclerosis. 2015 Jun;240(2):520-5. doi: 10.1016/j.atherosclerosis.2015.04.793. Epub 2015 Apr 22. PMID 25932792
- [Derived] Shearer GC, Pottala JV, Hansen SN, Brandenburg V, Harris WS. Effects of prescription niacin and omega-3 fatty acids on lipids and vascular function in metabolic syndrome: a randomized controlled trial. J Lipid Res. 2012 Nov;53(11):2429-35. doi: 10.1194/jlr.P022392. Epub 2012 Aug 14. PMID 22892157
- [Derived] Hu S, Shearer GC, Steffes MW, Harris WS, Bostom AG. Once-daily extended-release niacin lowers serum phosphorus concentrations in patients with metabolic syndrome dyslipidemia. Am J Kidney Dis. 2011 Jan;57(1):181-2. doi: 10.1053/j.ajkd.2010.06.029. Epub 2010 Oct 8. No abstract available. PMID 20888102
- See also: Abstract to Published Paper — http://www.ncbi.nlm.nih.gov/pubmed/22892157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from throughout the Sanford Clinic - Clinical Research Services in Sioux Falls by posted advertisements in public places and at sponsored health fairs.
Pre-assignment Details: 68 subjects willing to participate and qualified were subjected to a 6 week single blind run in period where they were given placebo omega-3 and placebo niacin. "Baseline" was defined as values and metrics after this run in period.
Groups:
- Dual Placebo: Dual placebo
  placebo: omacor placebo plus niaspan placebo
- Niaspan: niaspan
  extended release niacin: 2 g qpm
- Lovaza: lovaza
  omega-3 acid ethyl esters: 4 q qd
- Combined Therapy: combined therapy
  combined treatment: omega-3 acid ethyl esters 4 g qd and extended release niacin, titrate up to 2 g Qpm
Period: Overall Study
Arm/Group | Dual Placebo | Niaspan | Lovaza | Combined Therapy
Started | 17 | 17 | 17 | 17
Completed | 15 | 15 | 17 | 13
Not Completed | 2 | 2 | 0 | 4
Not completed — Protocol Violation | 1 | 2 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lovaza: lovaza
  omega-3 acid ethyl esters: 4 q qd
  omega-3 acid ethyl esters: 4 g qd
- Total: Total of all reporting groups
Arm/Group | Dual Placebo | Niaspan | Lovaza | Combined Therapy | Total
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 68
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [39 to 65] | 49 [41 to 56] | 44 [40 to 49] | 48 [44 to 54] | 46 [40 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 10 | 8 | 33
  Male | 10 | 9 | 7 | 9 | 35

OUTCOME MEASURES:

1. Primary Outcome: Serum TG
Description: Change From Baseline to 4 Months in Serum Triglycerides
Time Frame: 4 months
Population: Those subjects with complete data baseline to end
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dual Placebo | Niaspan | Lovaza | Combined Therapy
Number analyzed (Participants) | 15 | 15 | 17 | 13
mg/dl | 233 (162) | 157 (52) | 176 (63) | 156 (56)

2. Secondary Outcome: Non-HDL-C
Description: Change From Baseline to 4 Months in Serum Non-HDL cholesterol
Time Frame: baseline and 4 months
Population: all subjects with pre and post treatment data
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dual Placebo | Niaspan | Lovaza | Combined Therapy
Number analyzed (Participants) | 15 | 15 | 17 | 13
mg/dl | 145 (23) | 155 (43) | 133 (34) | 170 (36)

ADVERSE EVENTS:
Time Frame: 16 weeks of the intervention
Arm/Group | Dual Placebo | Niaspan | Lovaza | Combined Therapy
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/17 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No